CLINICAL TRIAL: NCT02733653
Title: A Prospective, Multicenter, Single-arm Clinical Trial of Jetstream Atherectomy System for the Treatment of Japanese Patients With Symptomatic Occlusive Atherosclerotic Lesions in the Superficial Femoral and/ or Proximal Popliteal Arteries
Brief Title: Safety and Effectiveness of Jetstream Atherectomy System (J-SUPREME)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6051
Record Dates: First submitted 2016-03-24; First posted 2016-04-11 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Peripheral Arterial Disease
Keywords: Superficial Femoral Artery; Proximal Popliteal Artery; Endovascular therapy; Atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Jetstream Atherectomy System (Experimental): Adjunctive therapy with Jetstream Atherectomy System for percutaneous intervention
  Interventions: Device: Jetstream Atherectomy System

INTERVENTIONS:
Device: Jetstream Atherectomy System — A rotating, aspirating, expandable catheter system for active removal of atherosclerotic debris and thrombus in the SFA and/or PPA

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Jetstream Atherectomy System for the treatment of Japanese patients with symptomatic occlusive atherosclerotic lesions in native superficial femoral artery (SFA) and/or proximal popliteal arteries (PPA).

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm trial evaluating the safety and efficacy of the Jetstream Atherectomy System in the treatment of symptomatic occlusive atherosclerotic lesions ≤150 mm in length located in the femoropopliteal arteries in subjects with symptoms classified as Rutherford categories 2-4.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2-4
* Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA of which meet all of the following criteria:

  * Calcified lesions with degree of stenosis ≥70% or occlusions
  * Guidewire must cross lesion(s) within the true lumen, without a sub-intimal course
  * Vessel diameter ≥3.0 mm and ≤6.0 mm
  * Total lesion length (or series of lesions) ≤150mm
  * Target lesion located at least 3 cm above the inferior edge of the femur by visual estimate
* Patent infrapopliteal and popliteal artery

Exclusion Criteria:

* Target lesion/vessel with in-stent restenosis
* Target lesion/vessel previously treated with drug-coated balloon <12 months prior to the procedure
* Target lesion/vessel previously treated with any stent placement, atherectomy, laser or other debulking devices prior to the procedure
* Subjects who have undergone surgery or endovascular of the SFA/PPA in the target vessel to treat atherosclerotic disease within 3 months prior to the index procedure
* Use of drug-coated devices, atherectomy, laser or other debulking devices other than the Jetstream System, chronic total occlusion (CTO) devices or cutting balloon, Angioscore or similar devices in the target limb SFA/PPA during the index procedure
* History of major amputation in the target limb
* Subject has a history of coagulopathy or hypercoagulable bleeding disorder
* Subject with untreatable hemorrhagic disease or platelet count <80,000mm3 or >600,000mm3 as baseline assessment.
* Concomitant renal failure with a serum creatinine >2.0 mg/dL
* Receiving dialysis or immunosuppressant therapy
* History of myocardial infarction, or stroke/cerebrovascular accident (CVA) within 6 months prior to study enrollment
* Unstable angina pectoris at the time of the enrollment
* Septicemia at the time of enrollment
* Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure
* Presence of aneurysm in the target vessel
* Acute ischemia and/or acute thrombosis of the SFA/PPA prior to the index procedure
* Perforated vessel as evidenced by extravasation of contrast media prior to the index procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazushi Urasawa, MD, PhD, Principal Investigator — Tokeidai Memorial Hospital
Locations (10):
- Japan (10):
  - Nagoya Kyoritsu Hospital, Nagoya, Aichi-ken
  - Kokura Memorial Hospital, Kokura, Fukuoka
  - Iwaki Kyouritsu Hospital, Iwaki, Fukushima
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Miyazaki Medical Association Hospital, Miyazaki
  - Nagano Red Cross Hospital, Nagano

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty patients including 10 roll-in patients were enrolled in this trial. Roll-in patients are not included in the endpoint analyses.
Groups:
- Jetstream Atherectomy System - Primary Subject: Adjunctive therapy with Jetstream Atherectomy System for percutaneous intervention
  Jetstream Atherectomy System: A rotating, aspirating, expandable catheter system for active removal of atherosclerotic debris and thrombus in the SFA and/or PPA
Period: Overall Study
Arm/Group | Jetstream Atherectomy System - Primary Subject
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Jetstream Atherectomy System - Primary Subject
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 72.3 [50.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 50
Region of Enrollment [Number; unit: participants]
  Japan | 50

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency Rate
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System - Primary Subject
Number analyzed (Participants) | 47
Participants | 19

2. Other Pre Specified Outcome: Procedural Success Rate
Description: Bailout stenting or surgical procedure during the index procedure is not needed
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System - Primary Subject
Number analyzed (Participants) | 50
Participants | 50

3. Other Pre Specified Outcome: Rate of Distal Emboli Requiring Additional Treatment
Time Frame: during procedure or within 24 hours post-index procedure
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Reduction in Lesion Stenosis
Description: The difference between the percent stenosis prior to treatment with Jetstream and the percent stenosis following treatment with Jetstream.
Time Frame: during procedure
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Major Adverse Event (MAE) Rate
Description: All-cause death through 1 month, and/or target limb major amputation and/or Target Lesion Revascularization (TLR) through 12 months
Time Frame: 1 month, 6 months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System - Primary Subject
Number analyzed (Participants) | 49
Participants
  MAE at 6 months | 5
  MAE at 12 months | 13

6. Other Pre Specified Outcome: Primary Patency
Description: Percentage (%) of lesions that reach endpoint without a hemodynamically significant stenosis on Duplex Ultrasound (DUS) and without Target Lesion Revascularization (TLR) or, bypass of the target lesion.
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assisted Primary Patency
Description: Percentage (%) of lesions without TLR and those with TLR (not due to complete occlusion or by-pass) that reach endpoint without restenosis.
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clinically-driven TLR Rate
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Clinically-driven Target Vessel Revascularization (TVR) Rate
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Adverse Event Rates
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Distribution of Rutherford Class
Description: Distribution of Rutherford Class as compared to baseline at 6 months and 12 months
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Rate of Primary and Secondary Sustained Clinical Improvement
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Rate of Hemodynamic Improvement
Time Frame: 1 month, 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Jetstream Atherectomy System - Primary Subject
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 25/50
Other Adverse Events (participants affected / at risk) | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Jetstream Atherectomy System - Primary Subject (N=50)
Peripheral artery occlusion (Vascular disorders) | 6
Peripheral artery stenosis (Vascular disorders) | 8
Arterial intramural haematoma (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Angina pectoris (Cardiac disorders) | 5
Acute myocardial infarction (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Jetstream Atherectomy System - Primary Subject (N=50)
Peripheral artery stenosis (Vascular disorders) | 11
Peripheral embolism (Vascular disorders) | 3
Nasopharyngitis (Infections and infestations) | 7
Vascular procedure complication (Injury, poisoning and procedural complications) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction depends on the conditions on the Clinical Study Agreement at each site. The PI must notify the sponsor about the publication and receive the approval from the sponsor prior to any results/data relavant to the J-SUPREME trial to be in public.

DOCUMENTS (2):
  • Study Protocol (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT02733653/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02733653/SAP_001.pdf